112406 (NYESO1-AS15-MEL-001 (MET) Statistical Analysis Plan Final

| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
|---|---|
| Detailed Title: | An open Phase I Study of immunization with the recNY-ESO-1 + AS15 Antigen-Specific Cancer Immunotherapeutic in patients with NY-ESO-1-positive unresectable and progressive metastatic cutaneous melanoma |
| eTrack study number and<br>Abbreviated Title | 112406 (NYESO1-AS15-MEL-001 (MET)) |
| Scope: | All data pertaining to the above study, with the exception of translational research analyses |
| Date of Statistical Analysis<br>Plan | Final 05-Apr-2018 |
| Co-ordinating author: | PPD |
| Reviewed by: | (Clinical Research and Development Lead) |
| | (SERM safety physician) |
| | PPD (SERM Scientist), |
| | (Scientific writer) |
| | (Lead Scientific writer) |
| | (Lead statistical analyst) |
| | (Public disclosure representative) |
| Approved by: | (Clinical and Epidemiology Project Lead) delegating to PPD (Clinical Research and Development Lead) |
| | (Lead statistical analyst) |
| | (Lead Scientific writer) |
| | (Lead statistician) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 14 April 2017)

112406 (NYESO1-AS15-MEL-001 (MET) Statistical Analysis Plan Final

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| LIS | T OF A | BBREVIA | ATIONS | 4 |
| 1. | DOC | JMENT H | IISTORY | 6 |
| 2. | STUE | N DESIG | iN | 6 |
| ۷. | 31001 DEGIGIN | | | |
| 3. | | | | |
| | 3.1.<br>3.2. | • | nary objectivesary objectives | |
| | | | • | |
| 4. | | | | |
| | 4.1. | | nary endpoints | |
| | | 4.1.1. | J 1 | |
| | 4.2. | 4.1.2. | Clinical activity endpoint | |
| | 4.2. | 4.2.1. | ary endpoints | |
| | | 4.2.1.<br>4.2.2. | Safety endpointsClinical activity endpoints | |
| | | 4.2.3. | Immunogenicity endpoints | |
| | | 7.2.0. | minunogeniony enapoints | |
| 5. | STUD | Y POPUI | LATION | 7 |
| | 5.1. | | eated population (TTP) | <mark>7</mark> |
| | 5.2. | | ng-to-protocol (ATP) population for analysis of | • |
| | | immund | ogenicity | 8 |
| 6. | STAT | ISTICAL | METHODS | 8 |
| | 6.1. | Screeni | ng | 8 |
| | 6.2. | | s of demographics/baseline characteristics | |
| | 6.3. | | ent exposure and compliance | |
| | 6.4. | | s of safety | |
| | 6.5. | | s of immunogenicity | |
| | 6.6. | Analysis | s of clinical activity | 10 |
| 7. | STAT | ISTICAL | CALCULATIONS | 11 |
| | 7.1. | | and transformed data | |
| | | 7.1.1. | Compliance | |
| | | 7.1.2. | Coding and Grading of Adverse events | |
| | | 7.1.3. | Humoral immune response to the administered recNY- | |
| | | | ESO-1 + AS15 ASCI | |
| | | 7.1.4. | Time-to-event calculation | |
| | | 7.1.5. | Last known alive date | |
| | 7.2. | Method | ology for computing CI | 13 |
| 8. | CON | DUCT OF | ANALYSES | 13 |
| | 8.1. | | ce of analyses | |
| | 8.2. | | cal considerations for interim analyses | |
| 9 | CHAN | IGES FR | OM PLANNED ANALYSES | 13 |

| 12406 (NYESO1-AS15-MEL-001 (MET) |
|----------------------------------|
| Statistical Analysis Plan Final |
| 14 |

## 112406 (NYESO1-AS15-MEL-001 (MET) Statistical Analysis Plan Final

#### **LIST OF ABBREVIATIONS**

AE Adverse event

ALT Alanine Aminotransferase

APTT Activated Partial Thromboplastin Time

AS GSK proprietary Adjuvant System (ex. AS01B, AS02B, AS07A...)

ASCI Antigen Specific Cancer Immunotherapeutic

AST Aspartate Aminotransferase

ATP According-To-Protocol

CD4 Cluster Differentiation marker-4 expressed by helper T-cells

CD8 Cluster Differentiation marker-8 expressed by cytotoxic T-cells

CI Confidence Interval

CR Complete Response

CMI Cellular Mediated Immunization

CTC Common Toxicity Criteria

CTCAE Common Terminological Criteria for Adverse Events

DSMC Data Safety Monitoring Committee

ECOG Eastern Cooperative Oncology Group

ELISA Enzyme-linked immunosorbent assay

GGT Gamma Glutamyl Transferase

GMC Geometric Mean antibody Concentration

GSK GlaxoSmithKline

MedDRA Medical Dictionary for Regulatory Activities

NE Non Evaluable

NSCLC Non-Small Cell Lung Cancer

PD Progressive Disease

112406 (NYESO1-AS15-MEL-001 (MET) Statistical Analysis Plan Final

PFS Progression Free Survival

PR Partial Response

SAE Serious Adverse Event

NY-ESO-1 Cancer-Testis gene: New York-ESOphageal cancer-1

SAP Statistical Analysis Plan

SD Stable Disease

SOC System Organ Class

TFL Tables Figures and Listing template annexed to SAP

TNM Tumor, Node, Metastasis (staging system for NSCLC)

TTF Time to Treatment Failure
TTP Total Treated Population

USA United States of America

112406 (NYESO1-AS15-MEL-001 (MET) Statistical Analysis Plan Final

## 1. DOCUMENT HISTORY

The SAP is divided into 2 parts: the first part detailing the analyses to be performed (current document) and a second part, annex (-es) (called TFL's) describing the flow and format of tables, figures and listings to be annexed to the SR

| Date | Version | Description | Protocol Version |
|-------------|---------------|----------------|-------------------------|
| 05-APR-2018 | Final version | Final analysis | Amendment 3 03-SEP-2014 |

#### 2. STUDY DESIGN

See protocol

The following group name will be used for the statistical analyses:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | Gr.1 | recNY-ESO-1 + AS15 ASCI |

#### 3. OBJECTIVES

# 3.1. Co-primary objectives

The two co-primary objectives of this study are to document and to characterize the severe toxicity and clinical activity of the recNY-ESO-1 + AS15 ASCI in patients with NY-ESO-1-positive metastatic cutaneous melanoma.

# 3.2. Secondary objectives

Note that, as of Amendment 3, the decision was taken not to perform further testing on biological samples already collected in this study by default, except if a scientific rationale remains relevant. No further blood samples for protocol research purposes will be collected.

The secondary objectives of this study are to document and characterize:

- 1. Additional clinical indicators of clinical activity in the overall population and in the population of patients who present the predictive MAGE-A3 gene signature\*.
- 2. Additional indicators of safety.
- 3. The specific humoral and cellular immune response\* induced by recNY-ESO-1 + AS15 ASCI.
  - \* changed from protocol (see section 9)

#### 4. ENDPOINTS

## 4.1. Co-primary endpoints

## 4.1.1. Safety endpoint

• Occurrence of severe toxicities during the study treatment phase and follow-up.

# 4.1.2. Clinical activity endpoint

• The induction of objective clinical response (CR or PR).

# 4.2. Secondary endpoints

## 4.2.1. Safety endpoints

• Occurrence of AEs and SAEs during the study treatment period and ending 30 days after the last study treatment administration.

## 4.2.2. Clinical activity endpoints

- Occurrence of stable disease (SD).
- Occurrence of mixed response (MR).
- Time to Treatment Failure (TTF).
- Progression-free survival (PFS).
- Overall survival (OS).
- The duration of response for patients with CR, PR or SD status.

## 4.2.3. Immunogenicity endpoints

- The anti-NY-ESO-1 humoral antibody concentration and response.
- The anti-NY-ESO-1 specific cellular (T-cell) response.\*

#### 5. STUDY POPULATION

# 5.1. Total treated population (TTP)

The total treated population will include all enrolled patients who have received at least one ASCI dose injection.

112406 (NYESO1-AS15-MEL-001 (MET) Statistical Analysis Plan Final

# 5.2. According-to-protocol (ATP) population for analysis of immunogenicity

Due to decision from ITx closure to prepare an abridged annex report, only TTP will be analyzed at final analysis. The ATP population for analysis of immunogenicity will thus be not applicable.

## 6. STATISTICAL METHODS

All statistical analyses will be performed using SAS version 9.3 under SAS Drug Development (SDD) version 4.3.

Unless otherwise specified, the different characteristics will be tabulated and analyzed by appropriate descriptive statistics:

- Frequency tables will be generated for categorical variables such as center.
- Mean, median, standard error will be provided for continuous data such as age.

## 6.1. Screening

The following summaries will be presented on the total screened population:

- Number of patients who are NY-ESO-1 positive screening failures and reasons of screening failure
- NY-ESO-1 expression test results: positive, negative, non-conclusive, missing
- NY-ESO-1 quantitative expression

## 6.2. Analysis of demographics/baseline characteristics

The following demographic (age, gender, etc.) and other baseline characteristics will be presented:

- Number of patients by country and by center
- Demographic characteristics: age, gender, geographic ancestry
- Disease characteristics: T, N, M categories, stage
- Primary tumor characteristics

112406 (NYESO1-AS15-MEL-001 (MET) Statistical Analysis Plan Final

## 6.3. Treatment exposure and compliance

The following summaries will be presented on the total treated population:

- Number and percentage of patients who received study treatment doses
- Reason for premature treatment discontinuation
- Listings of (serious) adverse events leading to treatment discontinuation and to study discontinuation
- Number of patients still on treatment at each planned visit of the treatment phase and list of withdrawn patients
- Reason for premature study discontinuation
- Number of patients still on study at each planned visit and list of withdrawn patients

# 6.4. Analysis of safety

The following summaries will be presented on the total treated population:

- List of patients with at least one severe toxicity as assessed by the investigator, and details of related AE/SAE
- Summary of all adverse events, by MedDRA System Organ Class and Preferred Term and by worst grade (within 31 days post treatment and all)
- Summary of all adverse events that are causally related to treatment administration, by MedDRA System Organ Class and Preferred Term and by worst grade
- Summary of (potential) immune-mediated disorders by worst grade
- Summary of (potential) immune-mediated disorders that are causally related to treatment administration, by worst grade
- Summary of all serious adverse events, by MedDRA System Organ Class and Preferred Term and by worst grade
- Summary of all serious adverse events that are causally related to treatment administration, by MedDRA System Organ Class and Preferred Term and by worst grade
- Listings of all SAEs
- Summary of on-study laboratory data by worst grade versus baseline grade
- Performance status: worst value on study versus baseline

112406 (NYESO1-AS15-MEL-001 (MET) Statistical Analysis Plan Final

# 6.5. Analysis of immunogenicity

The analyses will only be produced on the total treated population.

The following summaries will be presented:

- Anti- NY-ESO-1 antibody seropositivity rates and geometric mean concentration with 95% CIs by timepoint.
- Anti- NY-ESO-1 responses by timepoint.
- Reverse Cumulative Curve of anti- NY-ESO-1 antibody concentration at visit 5, 11 and 15
- Individual patient kinetic: anti- NY-ESO-1 antibody concentration (log scale) versus elapsed time since first dose
- Graph of the anti- NY-ESO-1 GMCs by timepoints.

# 6.6. Analysis of clinical activity

The following summaries will be presented on the total treated population:

- Best overall response per patient (categories: CR, PR, SD, SD/PR, PD, NE) :number and proportion of subjects falling into each category
- Overall clinical response rate: number of patients whose best overall response is PR or CR, divided by the total number of patients.
- Disease control rate: number of patients whose best overall response is: any CR, PR, SD or SD/PR, divided by the total number of patients.
- Proportion of patients who present a slow progressive disease and mixed response during the course of treatment
- Kaplan-Meier curves for Follow-up duration: time from the date of first ASCI to the date the patient was last known to be alive. Patients who died during the study will be censored on the date of death.
- Kaplan-Meier curves for TTF: time from the date of first ASCI to the date of last treatment administration for patients who discontinued the treatment prematurely, regardless of the reason for study treatment discontinuation. Patients who completed their full treatment phase or who are still on treatment at the time of analysis will be censored on their last study treatment administration date.
- Kaplan-Meier curves for PFS: time from the date of first ASCI to either the date of
  progressive disease (PD) or the date of death (regardless of the reason), whichever
  occurs first. Patients who were still alive at the time of analysis and without any
  documented disease progression are censored at the date of their last tumor
  assessment

112406 (NYESO1-AS15-MEL-001 (MET) Statistical Analysis Plan Final

• Kaplan-Meier curves for OS: time from the date of first ASCI to the date of death (regardless of the reason). Patients who were still alive at the time of analysis are censored at the last known alive date.

#### 7. STATISTICAL CALCULATIONS

#### 7.1. Derived and transformed data

## 7.1.1. Compliance

Permitted deviations from the stipulated date of visit (due, e.g. to week-ends or public holidays) are as follows:

- Cycle 1 (Doses 1 to 6):  $\pm$  3 calendar days
- Cycle 2 (Doses 7 to 12):  $\pm$  3 calendar days
- Cycle 3 (Doses 13 to 16):  $\pm$  4 calendar days
- Cycle 4 (Doses 17 to 24):  $\pm$  7 calendar days

#### 7.1.2. Coding and Grading of Adverse events

- Adverse events and serious adverse events are coded according to the MedDRA dictionary (at the level of System Organ Class and Preferred Term) based on the verbatim reports. This coding is made by a medically qualified person experienced in the company-specific coding conventions. The latest available dictionary version at the time of analysis will be used.
- Adverse events and laboratory tests are graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
- Patients who did not report any particular event will be considered as patients not experiencing this event.

# 7.1.3. Humoral immune response to the administered recNY-ESO-1 + AS15 ASCI

- Anti-NY-ESO-1 antibody ELISA assay cut-off: 179 ELU/mL.
- A seropositive patient is a patient whose anti-NY-ESO-1 antibody titer is greater than or equal to the cut-off value.
- Seroconversion in a patient is defined by the increase in anti-NY-ESO-1 antibodies from a titer below the cut-off level before the treatment to a titer above the cut-off level following treatment.

112406 (NYESO1-AS15-MEL-001 (MET) Statistical Analysis Plan Final

• A humoral response is defined as:

<u>For an initially seronegative patient</u>: an increase in the anti-NY-ESO-1 antibody titer to above the cut-off level (i.e seroconversion).

<u>For an initially seropositive patient</u>: an increase in anti-NY-ESO-1 antibody titer to a level at least two times higher than the pre-treatment titer.

- The geometric mean concentration (GMC) is calculated by taking the anti-logarithm of the mean of the log10 concentration transformations. Antibody concentration below the assay cut-off will be given an arbitrary value of half of the cut-off for the purpose of the calculation.
- For a given patient and given immunogenicity measurement, results of missing or non-evaluable measurements will not be replaced. Therefore, an analysis will exclude patients with missing or non-evaluable measurements.
- For the analysis performed on the total treated population, patients without immunogenicity measurements after ASCI treatment will be treated as nonresponders.

#### 7.1.4. Time-to-event calculation

The baseline reference date is defined as the date of first treatment.

In instances where periods between two dates are to be calculated (time-to-event endpoints), the convention to be used is as follows:

```
[later date] – [earlier date] + 1 day.
```

Should the result of this calculation be lower than 1, the time-to-event value will be re-set to 1 (event on Day 1) for the purpose of including the patient in the analysis.

When converting a number of days to other units, the following conversion factors will be used:

1 year = 365.25 days

1 month = 30.4375 days.

#### 7.1.5. Last known alive date

For each patient who is still alive at the time of analysis, a date the patient was last known to be alive (Last Known Alive - LKA - date) will be determined.

The date the patient was last known to be alive will be derived as the latest of the following dates: dates of visits/vaccinations, last contact dates, phone contact dates, laboratory assessment dates, tumor assessment dates, (S)AEs onset/resolution dates.

# 7.2. Methodology for computing CI

- The 95% CI for GMC is obtained by first computing the 95% CI for the mean of log10-transformed concentration assuming that they are normally distributed with unknown variance. The 95% CI for the GMC is then obtained by applying the reverse operation (10x) on the 95% CI for the mean of log10-transformed concentration.
- The exact 95% CIs of the seropositivity and response rates are calculated using Clopper-Pearson's exact method.
- Two-sided 95% confidence intervals for the median Time to Event will be computed by the Brookmeyer and Crowley method.

#### 8. CONDUCT OF ANALYSES

## 8.1. Sequence of analyses

| Description | Analysis<br>ID | Disclosure Purpose (CTRS=public posting, SR=study report, internal) | Dry run<br>review<br>needed (Y/N) | Study Headline Summary (SHS)requiring expedited communication to upper management (Yes/No) | Reference for<br>TFL |
|---|---|---|---|---|---|
| Final analysis | E1_01 | Abridged CSR and CTRS | N | N | TFL FA E1_01 |

# 8.2. Statistical considerations for interim analyses

Not applicable.

#### 9. CHANGES FROM PLANNED ANALYSES

- Following MAGRIT study (A double-blind, randomized, placebo-controlled Phase III study to assess the efficacy of recMAGE-A3 + AS15 Antigen-Specific Cancer immunotherapeutic as adjuvant therapy in patients with resected MAGE-A3-positive Non-Small Cell Lung Cancer) showed the absence of treatment effect in any of the primary, secondary, or exploratory analyses, clinical activity will not be reported within the population of patients who present the predictive MAGE-A3 gene signature.
- Cellular (T-cell) response will not be summarized as results only available for few patients
- Due to decision from ITx closure to prepare an abridged annex report, only TTP will be analyzed at final analysis.

112406 (NYESO1-AS15-MEL-001 (MET) Statistical Analysis Plan Final

# 10. REFERENCES

Brookmeyer, R., and Crowley, J. A Confidence Interval for the Median Survival Time. *Biometrics*, 38, 29–41, 1982.

Clopper, CJ and Pearson, ES. The use of confidence or fiducial limits illustrated in the case of the binomial. *Biometrika* 26: 404-413, 1934.

Kaplan, E. L. and Meier, P. "Nonparametric Estimation from Incomplete Observations," *Journal of the American Statistical Association*, 53, 457-481, 1958.